CLINICAL TRIAL: NCT05847465
Title: Study of Thermoregulation in Exercise Heat Stroke in the Military Environment
Acronym: EXPLO-MITO
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PBMD03-1; 2023-A00156-39 (Other: IDRCB)
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Heat Stroke
Keywords: Heat tolerance test
MeSH Terms: conditions — Heat Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Several biological samples will be collected:
  * Blood samples: 3 blood samples will be collected before Heat Tolerance Test (HTT), immediately after HTT, and 1 hour after HTT.
  * Sweat sample: A single sweat sample will be collected at the end of the HTT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group (exercise heat stroke patients): Participants enrolled in the case group have been experiencing exercise heat stroke and are participating in the main EXPLO-CCE study.
  Interventions: Other: Bike stress test; Other: Heat Tolerance Test; Other: Heat nociception test
- Control group (healthy individuals): Participants enrolled in the control group are healthy individuals who are participating in the main EXPLO-CCE study.
  Interventions: Other: Bike stress test; Other: Heat Tolerance Test; Other: Heat nociception test

INTERVENTIONS:
Other: Bike stress test — This is an incremental exercise under maximal pedaling on an Excalibur® type bike with electromagnetic brake over 36 minutes during which gas exchanges are continuously measured through a face mask (Cosmed®).
Other: Heat Tolerance Test — The test consists of a walk on a treadmill in shorts, bare chest or bra for women, at 5 km/h and 2% slope in an environment at 40°C, 40% relative humidity, without convection.
  During the test, rectal temperature, heart rate and skin temperature will be monitored continuously.
  The blood pressure will be measured manually every 30 minutes during the test.
Other: Heat nociception test — This test consists in applying a thermal flux generated by an infrared light source on a beam of 1 cm diameter on 2 areas of the dominant lower limb (glabrous face of the forearm and thenar eminence).
  Participants will be instructed to remove their limb as soon as the sensation of heat begins to become uncomfortable.
  The time between the beginning of the stimulus and the moment of withdrawal will be recorded.

SUMMARY:
The EXPLO-MITO study is an ancillary study from the main EXPLO-CCE study (NCT04593316; IDRCB: 2020-A01967-32).

The Heat Tolerance Test (HTT) is a physiological exploration that has several advantages for use in research and clinical settings. Unlike the walk-run test, it is performed under controlled conditions, both environmentally (temperature control, humidity, etc.) and in terms of effort intensity. In addition, there are published interpretation criteria for this test allowing to characterize thermoregulation profiles and to distinguish between Heat Intolerant (HI) and Heat Tolerant (HT) patients.

The reproducibility of this test and its performance in a climatic chamber allows a true comparison of thermophysiological responses (heart rate, rectal and skin temperatures, skin blood flow and sweat loss), which was not possible with the run-walk test, which was more a field test validating a physical aptitude for recovery (so-called "occupational" test) than a physiological exploration evaluating a response to stress by comparing it with the expected response in a population of young, healthy, properly trained subjects. Moreover, the HTT is a much less physiologically demanding test than the 8-km run. The HTT, which corresponds to a 2-hour walk at 5 km/h with a 2% slope at 40°C and 40% relative humidity, is a so-called "compensable" thermal stress; that is, under these conditions of exercise and environment, when the individual has normal thermoregulatory capacities, a thermal equilibrium plateau is reached during the second hour, when the individual's thermolysis capacities make it possible to compensate for the production of heat by the exercise and the gain of heat related to the environment. On average, this plateau is between 38° and 39°C. This is clearly not the case with our experience of physiological monitoring of the 8-km walk-run which rarely allows a temperature plateau to be reached and is accompanied by a temperature rise constantly above 39°C. In addition to being performed in the laboratory, this test is therefore completely safe.

For all these reasons (reproducibility, relevance, predictive value of recurrence), this test has been used for more than 30 years by the Israeli army for the assessment of these cases of exercise heat stroke before their return to work. There is therefore a fair amount of published data and hindsight on the use and interest of this test. The Israeli test has the highest level of recommendation (Grade A) of all the other published heat tolerance tests. Also, the availability of a climatic chamber means that this test can now be proposed as one of the explorations available to clinicians who have to decide on the fitness of soldiers after exercise heat stroke.

ELIGIBILITY:
Inclusion Criteria:

* Be included in the main EXPLO-CCE study;
* Subject trained or re-trained at 2 aerobic sessions per week;
* At least 2 months from the exercise heat stroke experience

Exclusion Criteria:

* Subject with a current medication treatment (for the control group only),
* Subject with a contraindication to the ingestion of a thermal capsule, namely:

  * Weight less than 37 kg
  * Inflammatory, motor or obstructive disease of the digestive tract
  * History of digestive surgery
  * Participant requiring a CT or MRI scan prior to removal of the thermal capsule (scheduled scan)
  * Presence of an implantable electronic device (e.g. pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This ancillary study will involve a subgroup of participants included in the case group (exercise heat stroke) and the control group of the main EXPLO-CCE study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of heat intolerant individuals based on the Heat Tolerance Test | Through study completion (48 months)
  Classification of participants between Heat Intolerant (HI) and Heat Tolerant (HT) will be determined according to measured rectal temperature.
  Participants will be classified as HI if they have at least one of the following criteria at HTT:
  * Rectal temperature > 38.5°C at the end of the 2 hours
  * Rectal temperature change during the second hour > 0.45°C

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided